CLINICAL TRIAL: NCT00752648
Title: A Phase I, Open-label, 3-way Crossover Trial in Healthy Subjects to Compare the Bioavailability of a Single Oral Dose of TMC435350 Formulated as 2 Different Solid Formulations to That of a Single Oral Dose of TMC435350 Formulated as a Powder Blend Capsule.
Brief Title: TMC435350-TiDP16-C106: A Phase I Trial to Compare the Bioavailability and Plasma Pharmacokinetics After a Single Oral Dose of TMC435350 of 2 Different Solid Formulations Relative to a Powder Blend Capsule
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tibotec Pharmaceuticals, Ireland (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR015415
Record Dates: First submitted 2008-09-11; First posted 2008-09-15 (Estimated); Last update posted 2010-04-28 (Estimated); Status verified 2010-04

CONDITIONS: Hepatitis C; HCV
Keywords: TMC435350-TiDP16-C106; TMC435350-C106; Bioavailability; Pharmacokinetics
MeSH Terms: conditions — Hepatitis C | interventions — Simeprevir

INTERVENTIONS:
Drug: TMC435350

SUMMARY:
The objectives are: to compare the oral bioavailability and plasma pharmacokinetics of TMC435350 for 2 different solid formulations to those of TMC435350 formulated as a powder blend in a capsule, after a single oral dose of 200 mg in healthy volunteers; to determine the short term safety and tolerability of TMC435350 after a single oral dose of 200 mg formulated in capsules with 2 different formulations and as a tablet in healthy volunteers

DETAILED DESCRIPTION:
This is a Phase I, open-label, 3-way crossover trial in 12 healthy adult volunteers to compare the oral bioavailability of a single 200 mg intake of TMC435350 salt, formulated as 2 different solid formulations (a tablet and a capsule) to that of a single 200 mg intake of TMC435350 salt, formulated as a powder blend in a capsule. TMC435350 is a protease inhibitor in development for treatment of chronic hepatitis C virus (HCV) infection. During 3 sessions, each volunteer will receive 3 treatments according to a classical 6-sequence, 3-period Williams design.The treatments administered are: Treatment A: single dose of 200 mg TMC435350 salt, formulated as a powder blend filled in a capsule. Treatment B: single dose of 200 mg TMC435350 salt, formulated in a tablet. Treatment C: single dose of 200 mg. MC435350 salt, formulated in beads filled in a capsule. All medication intakes will be oral and under fed conditions. There will be a washout period of at least 7 days between medication intakes in subsequent treatment sessions. Full pharmacokinetic profiles of TMC435350 will be determined up to 72 hours after administration in each session. Safety and tolerability will be monitored continuously throughout the trial. Treatments A, B and C: TMC435350 200mg on Day 1 of each session.Intakes will be oral and in fed conditions.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoking for at least 3 months prior to selection
* Normal weight as defined by a body mass index (BMI, weight in kg divided by the square of height in meters) of 18.0 to 30.0 kg/m2, extremes included
* Informed Consent Form (ICF) signed voluntarily before the first trial-related activity
* Able to comply with protocol requirements
* Normal 12-lead electrocardiogram (ECG) (in triplicate) at screening including: Normal sinus rhythm (heart rate [HR] between 40 and 100 bpm), QTc interval = 450 ms, QRS interval < 120 ms, PR interval = 220 ms
* Healthy on the basis of a medical evaluation that reveals the absence of any clinically relevant abnormality and includes a physical examination, medical history, vital signs, and the results of blood biochemistry, and hematology tests and a urinalysis carried out at screening.

Exclusion Criteria:

* Past history of heart arrhythmias (extrasystolic, tachycardia at rest) or having baseline prolongation of QTc interval > 450 ms, history of risk factors for Torsade de Pointes syndrome (hypokalemia, family history of long QT syndrome)
* Female, except if postmenopausal since more than 2 years, or posthysterectomy, or post-tubal ligation (without reversal operation)
* Hepatitis A, B, or C infection, or human immunodeficiency virus - type 1 (HIV-1) or HIV-2 infection at screening
* A positive urine drug test at screening. Urine will be tested to check the current use of amphetamines, benzodiazepines, cocaine, cannabinoids, and opioids
* Currently active or underlying gastrointestinal, cardiovascular, neurologic, psychiatric, metabolic, renal, hepatic, respiratory, inflammatory, or infectious disease
* Any history of significant skin disease such as, but not limited to, rash or eruptions, drug allergies, food allergy, dermatitis, eczema, psoriasis, or urticaria
* History of drug allergy such as, but not limited to, sulfonamides and penicillins, or drug allergy witnessed in previous trials with experimental drugs
* Participation in an investigational drug trial within 60 days prior to the first intake of trial medication.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2008-07; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
To compare the oral bioavailability and plasma pharmacokinetics of TMC435350 for 2 different solid formulations to those of TMC435350 formulated as a powder blend in a capsule, after a single oral dose of 200 mg in healthy volunteers;

SECONDARY OUTCOMES:
To determine the short term safety and tolerability of TMC435350 after a single oral dose of 200 mg formulated as capsules of 2 different formulations and as a tablet in healthy volunteers.

CONTACTS AND LOCATIONS:
Overall Officials: Tibotec Pharmaceuticals Limited Clinical Trial, Study Director — Tibotec Pharmaceutical Limited